CLINICAL TRIAL: NCT05621993
Title: Efficacy and Safety of Azvudine in the Treatment of Patients With Corona Virus Disease (COVID-19) Pneumonia in China: an Multi-center Observational, Ambispective Cohort, Real-world Study
Brief Title: An Observational, Ambispective Cohort Study of Azvudine in the Treatment of Patients With COVID-19 Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Qian Qi, Department of Respiratory, The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital, Qianfoshan Hospital
Other Study IDs: 2022-11-16-QFS
Record Dates: First submitted 2022-11-16; First posted 2022-11-18 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: COVID-19 Respiratory Infection
MeSH Terms: interventions — azvudine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Combination therapy group: Patients who are treated with the combination therapy of Azvudine and Chinese herbal medicine will be included in this group. The combination therapy is Azvudine treatment (5 mg once a day) within 48 hours of first positive nucleic acid testing for COVID-19, combined with Chinese herbal medicine treatment.
  Interventions: Drug: Azvudine
- Sequential therapy group: Patients who are treated with the sequential therapy of Azvudine and Chinese herbal medicine will be included in this group. The sequential therapy is Azvudine treatment (5 mg once a day) after 48 hours of first positive nucleic acid testing for COVID-19, combined with Chinese herbal medicine treatment.
  Interventions: Drug: Azvudine
- Non-standard therapy group: Patients are treated with Azvudine combined with Chinese herbal medicine treatment. But Azvudine treatment is discontinued before the nucleic acid turns negative.
  Interventions: Drug: Azvudine
- The control group: Patients are treated with Chinese herbal medicine without Azvudine.

INTERVENTIONS:
Drug: Azvudine — Azvudine is a small molecular antiviral drug. On August 9, 2022, Azvudine was included in the Diagnostic and therapeutic protocol for COVID-9 in China.
  Groups: Combination therapy group; Non-standard therapy group; Sequential therapy group

SUMMARY:
This is a multicenter, ambispective observational cohort study. The patients with corona virus disease 2019 (COVID-19) will be included in the study. The patients will be divided into 4 groups according to the treatment mode (Azvudine treatment group within 48 hours after the first positive for nucleic acid, Azvudine treatment group after 48 hours after the first positive for nucleic acid, short course of Azvudine treatment without nucleic acid turning negative, and the control group) . This study aims to analyze the efficacy and safety of Azvudine in the treatment of patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of COVID-19 pneumonia
* Patients with the ability to take medication orally

Exclusion Criteria:

* Severe vomiting and difficulty in taking oral medication or ingestion of drugs after oral administration
* Suspected or confirmed active systemic infection other than COVID-19 pneumonia
* Pregnant or lactating women
* Patients with mental disorders
* Patients with severe liver damage
* Patients who are treated with small molecule drugs such as Nirmatrelvir Tablets/Ritonavir Tablets(co-packaged)
* Patients who are treated with RNA-dependent RNA polymerase (RDRP) inhibitors (Junshipharma VV116, Ascletis Pharma Inc. Asc10, Kexing biopharm Shen26, and Molnupiravir).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients who were diagnosed as COVID-19 pneumonia will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2023-11-16 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Time from positive nucleic acid to negative | every 3 days
  The time from the day when patients are first positive nucleic acid to the day when the Ct value of nucleic acid test is ≥35 or the result of nucleic acid test is negative.

SECONDARY OUTCOMES:
Proportion of patients with relapsed positive nucleic acid test within 28 days after negative | up tp 28 days
Proportion of patients with adverse events | up tp 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Respiratory, The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital, #16766, Jingshi Road, Jinan City, Shandong Province, China, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No